CLINICAL TRIAL: NCT06244771
Title: An Open-Label, Phase 1/2 Dose Escalation, Dose Expansion and Cohort Expansion Study Evaluating the Safety, PK and Clinical Activity of FMC-376 in Participants With KRAS G12C Mutated Locally Advanced Unresectable or Metastatic Solid Tumors
Brief Title: A Study Evaluating FMC-376 in Participants With KRAS G12C Mutated Solid Tumors
Acronym: PROSPER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Frontier Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FMC-376-CL101
Record Dates: First submitted 2024-01-19; First posted 2024-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors With KRAS G12C Mutations; Solid Tumor, Adult; Unresectable Solid Tumor; Metastatic Solid Tumor; Non Small Cell Lung Cancer; Colorectal Cancer; KRAS G12C; Pancreatic Cancer
Keywords: Lung Cancer; KRAS; G12C
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1A: sequential; Phase 1B and Phase 2: parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMC-376 (Experimental): Dose Escalation, Dose Expansion, and Cohort Expansion; Administered for 21-day cycle
  Interventions: Drug: FMC-376

INTERVENTIONS:
Drug: FMC-376 — Oral Capsule

SUMMARY:
The goal of this clinical trial is to evaluate FMC-376 in participants with advanced solid tumors with KRAS G12C mutations. This clinical trial will be conducted in 3 parts: Phase 1A (Dose Escalation), Phase 1B (Dose Expansion), and Phase 2 (Cohort Expansion). Multiple dose levels in participants with advanced solid tumors will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumors with KRAS G12C mutation
* Received and progressed or been intolerant to prior standard therapy OR standard therapy is considered inappropriate OR an investigational agent is considered standard of care
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematological, renal, and hepatic function
* Agrees not to participate in another interventional study while receiving study drug

Exclusion Criteria:

* Leptomeningeal disease or carcinomatous meningitis
* Clinically significant toxicity resulting from prior cancer therapies
* Known or suspected hypersensitivity to FMC-376 or any components of the study drug
* Condition that would interfere with study drug absorption
* Any illness or medical history that would impact safety or compliance with study requirements or impact ability to interpret study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | Up to 21 Days
  Number of participants with Dose Limiting Toxicities (DLTs)
Adverse Events (AEs) | Approximately 24 Months
  Number of participants with treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of FMC-376 | Approximately 24 Months
  Cmax
Time to Reach Maximum Blood Concentration (Tmax) of FMC-376 | Approximately 24 Months
  Tmax
Minimum Observed Plasma Concentration (Cmin) of FMC-376 | Approximately 24 Months
  Cmin
Elimination Half-life (t1/2) of FMC-376 | Approximately 24 Months
  t1/2
Area Under Blood Concentration-Time Curve (AUC) of FMC-376 | Approximately 24 Months
  AUC
Volume of Distribution (Vd) of FMC-376 | Approximately 24 Months
  Vd
Clearance (CL) of FMC-376 from Blood Plasma | Approximately 24 Months
  CL
Overall Response Rate (ORR) | Approximately 24 Months
  Assess per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of Response (DOR) | Approximately 24 Months
  Assess per RECIST v1.1
Disease Control Rate (DCR) | Approximately 24 Months
  Assess per RECIST v1.1
Progression-Free Survival (PFS) | Approximately 24 Months
  Assess per RECIST v1.1
Overall Survival (OS) | Approximately 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Lead, Study Director — Frontier Medicines Corporation
Locations (26):
- United States (15):
  - University of California San Diego (UC San Diego) Health - Jacobs Medical Center - Moores Cancer Center, La Jolla, California
  - University of California Irvine (UCI) - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California San Francisco (UCSF) - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Florida Cancer Specialists and Research Institute, Lake Mary, Florida
  - Northwest Cancer Centers, Dyer, Indiana
  - The University of Kansas Cancer Center, Fairway, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Community Clinical Trials, Kingwood, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - UT Health San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (6):
  - Macquarie University, Macquarie Park, New South Wales
  - Tasman Health Care, Southport, Queensland
  - Icon Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - GenesisCare North Adelaide, North Adelaide, South Australia
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- South Korea (5):
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Severance Hospital, Seoul, Seodaemun-gu
  - Korea University Anam Hospital, Seoul, Seongbuk-gu
  - Seoul National University Bundang Hospital, Gyeonggi-do, Seongnam-si
  - The Catholic University of Korea, St. Vincent's Hospital, Gyeonggi-do, Suwon-si

IPD SHARING:
Plan to Share IPD: No